CLINICAL TRIAL: NCT06277674
Title: A Phase II Clinical Trial Evaluating the Efficacy of Cadonilimab in Combination With Pemetrexed and Anlotinib for Treatment of Elderly Patients With T790M-negative Advanced Non-squamous Non-small Cell Lung Cancer Following Resistance to EGFR-TKI.
Brief Title: Efficacy of Cadonilimab in Non-squamous Non-small Cell Lung Cancer Patients Resistant to EGFR-TKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Principal Investigator, Haibo Zhang, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZF2023-252
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Cadonilimab; Immune checkpoint inhibitors; EGFR-TKI resistance; elderly non-small cell lung cancer patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; anlotinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cadonilimab plus pemetrexed and anlotinib (Experimental): Twenty elderly patients (age≥65 years) with advanced non-squamous NSCLC with T790M negative after EGFR-TKI resistance will be enrollrd in this study. Participants will receive 4 to 6 cycles of cardunnilumab in combination with pemetrexed and anlotinib every 3 weeks, followed by maintenance treatment with cadonilimab plus anlotinib until disease progression, intolerable toxicity, withdrawal of consent, death, or other protocol-specified causes, whichever occurs first.
  Cadonilimab was administered intravenously at a dose of 10 mg/kg every 3 weeks. Pemetrexed was administered intravenously at a dose of 500 mg/m² every 3 weeks Anlotinib was taken at doses of 10mg orally once daily for two weeks on a one-week-off schedule.
  Interventions: Drug: Cadonilimab plus Pemetrexed and Anlotinib

INTERVENTIONS:
Drug: Cadonilimab plus Pemetrexed and Anlotinib — Cadonilimab was administered intravenously at a dose of 10 mg/kg every 3 weeks. Pemetrexed was administered intravenously at a dose of 500 mg/m² every 3 weeks Anlotinib was taken at doses of 10mg orally once daily for two weeks on a one-week-off schedule.
  Other Names: ICIs in combination with chemotherapy and antiangiogenic therapy

SUMMARY:
This study was designed to evaluate the efficacy and safety of cadonilimab (anti PD-1 and CTLA-4 bispecific antibody) in combination with pemetrexed and anlotinib for treatment of elderly patients with T790M-negative advanced non-squamous non-small cell lung cancer following resistance to EGFR-TKI.

DETAILED DESCRIPTION:
This prospective study aims to enroll 20 elderly patients (age≥65 years) with advanced non-squamous NSCLC with T790M negative after EGFR-TKI resistance. Eligible patients will be given 4 to 6 cycles of cadonilimab plus pemetrexed and anlotinib, followed by maintenance treatment with cadonilimab plus anlotinib until disease progression, intolerable toxicity, withdrawal of consent, death, or other protocol-specified causes, whichever occurs first. Imaging assessments are scheduled to conduct every 6 weeks for the first year and then every 12 weeks thereafter. The follow-up of participants who discontinued treatment for reasons unrelated to disease progression will be continued, until the initiation of other anti-tumor therapy, disease progression, death, or the end of the study, whichever occurrs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients signed informed consent, willing to accept this regimen, able to adhere to the medication, and had good compliance.
2. Patients with advanced or metastatic non-small cell lung cancer (stage IIIB, IIIC, or IV according to the AJCC staging system, 8th edition) diagnosed by histopathology or cytopathology
3. Histologically or cytologically confirmed, locally advanced or metastatic nonsquamous non-small-cell lung cancer (stage IIIB, IIIC, or IV according to the AJCC staging manual, 8th edition) patients with EGFR sensitive mutations (confirmed by tumour histology, cytology, or cell-free or circulating tumour DNA) progressed after receiving EGFR tyrosine-kinase inhibitor therapy; confirmed EGFR Thr790Met negative mutation status after receiving first-generation, second-generation or third-generation EGFR tyrosine-kinase inhibitor as first-line or second-line treatment
4. Eastern Cooperative Oncology Group performance status of 0 to 2
5. Presence of at least one measurable lesion
6. An estimated life expectancy of at least 3 months
7. Good organ function was defined as hemoglobin≥90g/L (no blood transfusion within 7 days), absolute neutrophil count ≥1.5×109/L, and platelet count≥100×109/L. Total bilirubin level≤1.5 times of the upper limit of normal value (ULN), albumin ≥30g/L, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times of upper limit of normal (ULN), in cases with liver metastasis, AST and ALT≤5 times of ULN; Creatinine ≤1.5 times of ULN; International normalized ratio (INR) or prothrombin time (PT) ≤1.5 times of ULN, if the participant is receiving anticoagulant therapy normally, as long as the PT is within the prescribed range of anticoagulant drugs

Exclusion Criteria:

1. Concomitant driver mutations for which there were known therapies were identified, including but not limited to ALK rearrangement, ROS1 fusion, or BRAF V600E mutation
2. Previously received systemic anti-tumour therapy (including cytotoxic chemotherapy and antiangiogenic therapy) except EGFR tyrosine-kinase inhibitors for advanced NSCLC
3. Previously received immunotherapy (including anti-PD-1, anti-PD-L1, or anti-CTLA-4) antibodies or agents
4. The presence of an active malignancy within 2 years prior to the first dose was not allowed. Participants with locally cured tumors, such as basal-cell carcinoma or squamous-cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the breast, were not excluded
5. The enrollment of another clinical study was excluded except for observational or noninterventional studies or interventional studies with a follow-up period exceeding four weeks after the last dose of the study drug or more than five half-lives of the study drug
6. Patients received systemic treatment with Chinese patent medicine or Chinese herbal medicine exhibiting anti-tumor properties or immunomodulatory drugs (such as thymosin, interferon, interleukin) indicated for anti-tumor purposes within a 2-week period prior to the initial dosage
7. Participants with an active, known, or suspected autoimmune disease or a history of autoimmune disease are excluded from the study, except for those with Vitiligo, alopecia, Graves' disease, psoriasis, or eczema that do not require systemic treatment for nearly 2 years. Additionally, Participants with asymptomatic hypothyroidism (due to autoimmune thyroiditis) or stable doses of hormone replacement therapy and type I diabetes requiring only stable doses of insulin replacement therapy are also exempted. Furthermore, participants who had childhood asthma that has completely resolved and no longer require any intervention in adulthood or whose disease does not recur without an external trigger are eligible for inclusion
8. Participants who have received systemic treatment with corticosteroids (prednisone equivalent dose > 10 mg/day) or other immunosuppressive drugs within 14 days prior to the first dose are excluded
9. Documented history of immunodeficiency
10. Documented history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
11. Major surgical procedures (such as laparotomy, thoracotomy, viscerectomy, etc.) or severe trauma within 28 days prior to the initial administration (intravenous drip replacement is acceptable); Surgery aimed at improving or reducing the risk of oncologic complications within 14 days before the first dose; Or incomplete recovery from any of the aforementioned previous surgeries. Major surgical procedures were planned (at the investigator's discretion) within 30 days after the initial dose. Local surgery (e.g., placement of systemic ports, core needle biopsy) was permitted if performed at least 24 hours prior to initiation of study treatment
12. Patients with a medical history of gastrointestinal perforation, gastrointestinal fistula, or female genital fistula (such as vesicovaginal fistula, urethrovaginal fistula, etc.) within the past 6 months prior to the initial drug administration were eligible for enrollment if the perforation or fistula had been surgically treated (e.g., excision or repair) and if complete recovery or resolution of the condition was confirmed by the investigator
13. The presence of interstitial lung disease, whether symptomatic or not, may hinder the detection or management of suspected drug-related pulmonary toxicity
14. The presence of active pulmonary tuberculosis (TB). Patients suspected to have active TB underwent examination through chest X-ray and sputum analysis, while being assessed for clinical signs and symptoms

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective response rate) | From date of randomization until the date of death or date of withdraw, whichever came first, assessed up to 120 months
  ORR (overall response rate) is defined as sum of complete response (CR) rate and partial response (PR) rate, according to RECIST v 1.1, based on the chest, abdomen and/or brain CT/MRI evaluation. Patients will undergo a follow-up imaging examination every 6 weeks for the first year and then every 12 weeks thereafter.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  The time from the date of randomization to the date of disease progression, date of withdraw, or death from any cause, whichever occurs first.
(Disease control rate assessed by investigators) DCR (CR+PR+SD) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  DCR (disease control rate) is defined as sum of complete response (CR) rate, partial response (PR) rate and stable disease (SD) rate, according to RECIST v 1.1, based on the chest, abdomen and/or brain CT/MRI evaluation. Patients will undergo a follow-up imaging examination every 6 weeks for the first year and then every 12 weeks thereafter.
Overall survival (OS) | From date of randomization to the date of withdraw or date of death from any cause, whichever occurs first, assessed up to 120 months.
  The time from the date of randomization to the date of withdraw or date of death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Prof, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No